CLINICAL TRIAL: NCT06740994
Title: Ultrasound Guided Midline Continuous Spinal Anesthesia in the Elderly : is There an Advantage Over Conventional Landmark Paramedian Technique: a Randomized Controlled Trial
Brief Title: Ultrasound Guided Midline vs Landmark Paramedian Continous Spinal Anesthesia in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Sameh Ben Ahmed, Associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTEM USSA
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Spinal Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paramedian landmark group (Experimental): conventional landmark paramedian approach will be performed. isobar bupivacaine will be injected for continuous spinal anesthesia.
  Interventions: Procedure: conventional landmark paramedian technique
- Midline ultrasound group (Active Comparator): preprocedural ultrasound guided midline approach will be performed. isobar bupivacaine will be injected for continuous spinal anesthesia.
  Interventions: Procedure: preprocedural ultrasound guided midline technique

INTERVENTIONS:
Procedure: conventional landmark paramedian technique — a blind landmark scanning will be done and skin marking of the best palpable spinous process will be made.
  the site of injection will be determined by palpation. continuous spinal anesthesia will be performed via paramedian approach.
  Other Names: PML
  Arms: paramedian landmark group
Procedure: preprocedural ultrasound guided midline technique — a preprocedural ultrasound scanning will be done, and skin marking of the best quality space will be made.
  the site of injection and the insertion angle of the needle will be determined by ultrasound.
  continuous spinal anesthesia will be performed via midline approach.
  Other Names: MUS
  Arms: Midline ultrasound group

SUMMARY:
Former clinical studies have reported the superiority of the landmark guided paramedian approach above the classical landmark guided midline approach for the continuous spinal anesthesia especially in the elderly. On the other hand, more recent clinical trials have suggested that the use of ultrasound to guide spinal anesthesia will be safer and more effective than the conventional palpation-guided technique.

The aim of this study will be to compare the conventional "blind" landmark paramedian approach to the ultrasound "modern" guided midline approach for the continuous spinal anesthesia in the elderly with hip fractures.

Patients will randomly divided into two groups:

Group(PML): will undergo conventional landmark guided paramedian continuous spinal anesthesia Group (MUS): will undergo ultrasound guided midline continuous spinal anesthesia

DETAILED DESCRIPTION:
All elderly patients above 65 years old scheduled for elective surgery for hip fracture under continuous spinal anesthesia will be included in the study.

Patients will randomly divided into two groups by using random number generating software (Research Randomizer Version 4.0) Group(PML): will undergo conventional landmark guided paramedian continuous spinal anesthesia Group(MUS) : will undergo ultrasound guided midline continuous spinal anesthesia A written informed consent will be obtained from all participants, who will be blinded as to their allocated group.

After establishing a baseline monitoring (3 lead ECG, pulse oximetry and non-invasive blood pressure) and an intravenous access, a fascia-iliaca ultrasound guided block at the fractured hip will be performed for all patients by the injection of 20 ml of 1.5 % lidocaine.

15 minutes later with the aid of an assistant, the patient will be positioned at the edge of the operating table in an arched back posture.

In both groups the continuous spinal anesthesia(CSA) will be performed with one of three anesthesiologists (two residents in their fourth year of training anesthesia and one associate professor), each have sufficient experience in performing neuraxial ultrasound scans prior to the study. To fulfill this they will use an 18 gauge Tuohy needle with a 22 gauge intrathecal catheter.

In group PML:

The anesthesiologist will star by drawing the 10th rib line then he will by palpation identify the most prominent spinous process beneath. At this level he will mark on the patient skin the point of injection which will be1 cm lateral and 1 cm caudal to the caudal edge of the spinous process chosen.

After infiltration of the skin with 3 ml of 1% lidocaine at the marked site, the anesthesiologist will introduce the tuohy needle in a cephalomedial direction 10 to 15° off the sagittal plane.

when cerebrospinal fluid will be obtained, the CSA (continuous spinal anesthesia) catheter will be advanced 3 cm cephalad to the intrathecal space and taped to the skin.

The patient will be then returned to dorsal position and a volume of 30 ug of fentanyl and 3 ml of 0.1% isobar bupivacaine will be injected intrathecally via the catheter.

The intervertebral level at which the injection will be done,will be scanned with ultrasound at the end of the surgery, before CSA catheter withdrawal.

In group MUS:

The anesthesiologist will use a portable ultrasonography with a curved 2-5 MHz (Mega Hertz) probe to detect the sacrum in the paramedian sagittal oblique view (PSO) of the neuroaxis.

Than the transducer will be moved cephalad to scan the quality of interspinous spaces from L5/S1 to L2/L3. The interlaminar space that will have the best PSO quality i.e the clearest and largest ultrasound image of the posterior complex ( ligamentum flavum and posterior dura) and anterior complex ( posterior longitudinal ligament and anterior dura) will be chosen as the interspace for injection.

At this level a skin marker will be used to mark the midpoint of the short borders of the probe. Following this the probe will be rotated by 90° to obtain the transverse median view (TM) and by the same way the midpoint of the short borders of the probe will be marked.

The intersection of these two marks will be used as the point of injection. Similarly skin will be infiltrated with lidocaine and the tuohy needle will be inserted in the cephalomedial plane with a cephalad angle estimated by the probe inclination in the TM view.In this group, the anesthesiologist will not palpate the landmarks except he changing technique.For the rest of the procedure, the same steps will be followed.

In both groups, an alternative technique would be used if unsuccessful after 3 attempts( landmark/ultrasound guided paramedian approach for MUS Group ; landmark/ultrasound midline approach for PML Group).

For all participants strict asepsis will be respected throughout all the procedure, The distance needed to reach the intrathecal space from the skin will be recorded and the quality of the interspinous spaces chosen will be noted in the PSO and TM ultrasound views using a predefined scale (good = both posterior and anterior complex visible ; intermediate = posterior or anterior complex visible ; poor = neither complex visible)

ELIGIBILITY:
Inclusion Criteria:

* all consented patients aged over 65 years old scheduled to undergo surgery for hip fracture under continuous spinal anesthesia with American Society of Anesthesiologists ASA physical status classification from I to III

Exclusion Criteria:

* contraindications to spinal anesthesia ( allergy to local anesthetic, coagulopathy, infection at the site of injection)
* previous history of lumbar spine surgery
* per operative severe complication with conversion to general anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
the difference in number of needle passes between the two groups | from the first insertion of the needle until the fixation of the continuous spinal anesthesia catheter to patient skin
  the number of forward advancements of the Tuohy needle in a given interspinous space (i.e withdrawal and redirection of Tuohy needle without exiting the skin)

SECONDARY OUTCOMES:
number of spinal needle insertion attempts | from the first insertion of the needle until the fixation of the continuous spinal anesthesia catheter to patient skin
  the number of times the tuohy needle was withdrawn from the skin and reinserted
the rate of first pass success | from the first insertion of the needle until the fixation of the continuous spinal anesthesia catheter to patient skin
  a single needle insertion with no redirection
time for identifying landmarks | time taken from start of palpating or ultrasound scanning to the marking of the needle entry point
  in group PML: time from which the anesthesiologist started palpating to identify the landmarks to the needle entry point marking in group MUS: time from which the ultrasound probe was placed on the skin to the needle entry point marking
time taken for performing continuous spinal anesthesia | time taken from the start of the first insertion of the needle to the completion of fixation of the catheter to patient skin
  time from first needle insertion to fixation of continuous spinal anesthesia catheter to patient skin
incidence of continuous spinal anesthesia complications | from the star of first needle insertion to the completion of the continuous spinal anesthesia
  defined as: incidence of radicular pain, parasthesia and blood in the Tuohy needle
the injection level | from the start of identifying landmarks until the patient leaves the operation room
  the interspinous level at which dural puncture was done

CONTACTS AND LOCATIONS:
Overall Officials: MECHAAL BEN ALI, Professor, Principal Investigator — university manar Tunis, Tunisia
Locations (1):
- BEN ALI MECHAAL, Professor, Nabeul, Mrazga, Tunisia